CLINICAL TRIAL: NCT06326463
Title: CAR T-cell Therapy Directed to CD70 for Pediatric Patients With Hematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIRECT70; NCI-2024-03240 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancy; ALL, Childhood; AML, Childhood; Lymphoma; MDS
MeSH Terms: conditions — Hematologic Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD70- CAR T cell Therapy (Experimental): Patients will receive autologous (their own) cells.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: CD70-CAR T cell infusion (Autologous); Drug: Mesna

INTERVENTIONS:
Drug: Fludarabine — 40mg/m2, Day -4, -3 and -2
  Other Names: Fludara
Drug: Cyclophosphamide — Day -3 and Day-2
  REST DAY, -1
  Other Names: Cytoxan
Drug: CD70-CAR T cell infusion (Autologous) — Day 0 or +1
Drug: Mesna — Mesna is generally dosed at approximately 25% of the cyclophosphamide dose. It is generally given intravenously prior to and again at 3, 6 and 9 hours following each dose of cyclophosphamide
  Other Names: Mesnex

SUMMARY:
The study participant has one of the following blood cancers: acute myelogenous leukemia (AML)/myelodysplastic syndrome (MDS), acute lymphoblastic leukemia (B-ALL, T-ALL) or Lymphoma. Your cancer has been difficult to treat (refractory) or has come back after treatment (relapse).

Primary Objective

To determine the safety and maximum tolerated dose of intravenous infusions of escalating doses of CD70-CAR T cells in patients (≤21 years) with recurrent/refractory CD70+ hematological malignancies after lymphodepleting chemotherapy.

Secondary Objectives

To evaluate the antileukemic activity of CD70-CAR T cells. We will determine the anti- leukemic activity of the CD70-CAR T cells in the bone marrow and in the treatment of extramedullary disease.

DETAILED DESCRIPTION:
The primary interventions are a lymphodepleting chemotherapy regimen (fludarabine and cyclophosphamide), followed by a single autologous infusion of CD70-CAR T cells.

Phase I study evaluating three (3) dose levels of CD70-CAR T cells.

ELIGIBILITY:
Inclusion Criteria

Age ≤21 years old

Relapsed/refractory CD70+ hematological malignancy

Relapsed disease: Patients developing recurrent disease after a prior complete remission (CR)

Refractory disease: Patients with persistent disease despite 3 cycles of induction chemotherapy.

* Relapsed/refractory CD70+ AML or MDS:

  * Relapsed disease that is CD70 positive
  * Refractory disease that is persistent despite 3 cycles of chemotherapy
* Relapsed/refractory CD70+ B-cell ALL:

  * Relapsed disease that is CD70 positive and CD19 negative/dim or patients otherwise ineligible for CD19-directed therapies including:
  * Patients in 2nd or greater relapse
  * Patients with relapse after allogeneic HSCT
* Relapsed/refractory CD70+ T-cell ALL:

  * Relapsed /refractory disease that is CD70 positive
* Mixed Phenotype Acute Leukemia (MPAL):

  * Relapsed/refractory that is CD70 positive
* Relapsed/refractory CD70+ lymphoma:

  * Relapsed disease that is CD70 positive and CD19 negative/dim or patients otherwise ineligible for CD19-directed therapies including:
  * Patients in 2nd or greater relapse
  * Patients with relapse after allogeneic HSCT

Estimated life expectancy of >12 weeks

Karnofsky or Lansky (age- dependent) performance score ≥50

Patients with a history of prior allogeneic HCT must be clinically recovered from prior HCT therapy, have no evidence of active GVHD and have not received a donor lymphocyte infusion (DLI) within the 28 days prior to apheresis

Patient must have an identified HCT donor

For females of childbearing age:

i. Not lactating with intent to breastfeed

ii. Not pregnant with negative serum or urine pregnancy test within 7 days prior to enrollment

Exclusion Criteria

* Known primary immunodeficiency
* Known history of HIV positivity
* Severe intercurrent bacterial, viral or fungal infection
* History of hypersensitivity to cornstarch or hydroxyethyl starch
* Patients with acute promyelocytic leukemia (APL)
* Known contraindication to protocol defined lymphodepleting
* chemotherapy regimen of Fludarabine/cyclophosphamide

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of CD70-CAR T cells | 28 days after CD70-CAR T-cell infusion
  Phase I design to determine the maximum tolerated dose (MTD) of autologous, CD70-CAR T cells. Three (3) dose levels will be evaluated (1x10e6, 3x10e6, and 1x10e7 cells/kg).

CONTACTS AND LOCATIONS:
Overall Officials: Swati Naik, MBBS, Principal Investigator — St. Jude
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols